CLINICAL TRIAL: NCT05169515
Title: A Phase Ib, Open-Label, Multicenter Study Evaluating the Safety, Pharmacokinetics, and Efficacy of Mosunetuzumab or Glofitamab in Combination With CC-220 and/or CC-99282 in Patients With B-Cell Non-Hodgkin Lymphoma
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Efficacy of Mosunetuzumab or Glofitamab in Combination With CC-220 and/or CC-99282 in Participants With B-Cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO43805
Record Dates: First submitted 2021-12-13; First posted 2021-12-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — glofitamab; iberdomide; obinutuzumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants will receive subcutaneous (SC) mosunetuzumab + CC-220 (dose escalation only) or SC mosunetuzumab + CC-99282.
  Interventions: Drug: SC Mosunetuzumab; Drug: Iberdomide; Drug: Golcadomide; Drug: Tocilizumab
- Arm 2 (Experimental): Participants will receive intravenous (IV) glofitamab + CC-99282.
  Interventions: Drug: IV Glofitamab; Drug: Golcadomide; Drug: Obinutuzumab; Drug: Tocilizumab

INTERVENTIONS:
Drug: SC Mosunetuzumab — Participants will receive SC mosunetuzumab for 12 cycles (cycle length = 21 days or 28 days for Cycle 1 and 28 days for Cycles 2-12)
  Other Names: RO7030816
  Arms: Arm 1
Drug: IV Glofitamab — Participants will receive IV glofitamab for 12 cycles (cycle length = 21 days)
  Other Names: RO7082859
  Arms: Arm 2
Drug: Iberdomide — Arm 1: Participants will receive oral CC-220 from Day 1-21 of Cycle 2-12 (cycle length = 28 days for Cycles 2-12)
  Other Names: CC-220
  Arms: Arm 1
Drug: Golcadomide — Arm 1: Participants will receive oral golcadomide from Day 1-14 starting in either Cycle 1 or Cycle 2 through Cycle 12 (cycle length = 28 days for cycles when golcadomide is to be administered) Arm 2: Participants will receive oral golcadomide from Day 1-10 starting in either Cycle 1, Cycle 2 or Cycle 3 through Cycle 12 (cycle length = 21 days)
  Other Names: CC-99282
Drug: Obinutuzumab — Participants in Arm 2 will receive pre-treatment with IV obinutuzumab on Cycle 1 Day 1 (cycle length = 21 days)
  Other Names: RO5072759
  Arms: Arm 2
Drug: Tocilizumab — Participants will receive IV tocilizumab as needed to manage cytokine release syndrome (CRS)
  Other Names: RO4877533

SUMMARY:
This study will evaluate the safety, efficacy, and pharmacokinetics of mosunetuzumab or glofitamab in combination with CELMoDs (CC-220 and/or CC-99282) in participants with B-cell NHL.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* History of one of the following histologically documented hematologic malignancies that are expected to express the CD20 antigen: In the Dose Escalation phase, participants must have relapsed after or failed to respond to at least two prior lines of systemic therapy. In the Dose Expansion phase, participants with FL Grades 1-3a must have relapsed after or failed to respond to at least one prior line of systemic therapy and must require systemic therapy. Participants with DLBCL/transformed FL must have relapsed after or failed to respond to at least one prior systemic treatment regimen.
* Participants with DLBCL/transformed FL who have received only one prior line of therapy must: Not be considered a candidate for autologous stem cell transplantation (ASCT) due to age, performance status, comorbidities and/or insufficient response to prior treatment, or have refused ASCT; or be ineligible for or unable to receive chimeric antigen receptor T-cell (CAR-T) therapy due to reasons defined by the protocol
* Fluorodeoxyglucose-avid lymphoma (i.e. PET-positive lymphoma)
* At least one bi-dimensionally measurable nodal lesion (> 1.5 cm in its largest dimension by diagnostic quality CT or PET/CT scan), or at least one bi-dimensionally measurable extranodal lesion (> 1.0 cm in its largest dimension by diagnostic quality CT or PET/CT scan)
* Availability of a representative tumor specimen and the corresponding pathology report for confirmation of the diagnosis of NHL
* A fresh pretreatment biopsy during screening period, excisional or incisional, is preferred
* Adequate hematologic function without growth factors or blood product transfusion within 14 days of first dose of study drug administration
* Normal laboratory values
* All participants and health care providers will be trained and counseled on pregnancy prevention. For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception during the treatment period and for 3 months after the final dose of mosunetuzumab, at least 18 months after pre-treatment with obinutuzumab or 2 months after the last dose of glofitamab, 28 days after the last dose of CC-220, 28 days after the last dose of CC-99282, 3 months after the last dose of tocilizumab (if applicable), whichever is longer
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agree to refrain from donating sperm during the treatment period and for at least 3 months after pre-treatment with obinutuzumab or 2 months after the last dose of glofitamab, 28 days after the last dose of CC-220, 28 days after the last dose of CC- 99282, 2 months after the final dose of tocilizumab (if applicable), whichever is longer

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention of becoming pregnant during the study (female participants of childbearing potential must have a negative serum pregancy test result within 14 days prior to initiation of the study treatment) or within 3 months after the final dose of mosunetuzumab, at least 3 months after pre-treatment with obinutuzumab or 2 months after the last dose of glofitamab, whichever is longer, 28 days after the last dose of CC-220, 28 days after the last dose of CC-9282, 3 months after the final dose of tocilizumab, whichever is longer
* Participant has received prior therapy with cereblon (CRBN)-modulating drug (e.g., lenalidomide, avadomide/CC-122, pomalidomide) </= 4 weeks prior to starting CC-220 and/or CC-99282
* Inability to swallow pills, or persistent diarrhea or malabsorption >= Grade 2 National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), despite medical management
* QTc interval of > 470 ms
* The following treatments prior to study entry: mosunetuzumab, glofitamab, or other CD20/CD3-directed bispecific antibodies; allogenic stem cell therapy (SCT); solid organ transplantation
* Treatments (investigational or approved) within the following time periods prior to initiation/first dose of study treatment: radiotherapy within 2 weeks; autologous SCT within 100 days; chimeric antigen receptor (CAR) T-cell therapy within 30 days; prior anti-lymphoma treatment with monoclonal antibodies or antibody-drug conjugates within 4 weeks; use of radioimmunoconjugates within 12 weeks; systemic immunosuppressive medications within 2 weeks; any other anti-cancer therapy, whether investigational or approved, including but not limited to chemotherapy, within 4 weeks or 5 half-lives of the drug, whichever is shorter
* Live, attenuated vaccine within 4 weeks before first dose of study treatment, or in whom it is anticipated that such a live attenuated vaccine will be required during the study period or within 5 months after the final dose of study treatment
* Current or past history of central nervous system (CNS) lymphoma or leptomeningeal infiltration
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* History of autoimmune disease, including but not limited to myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, granulomatosis with polyangiitis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
* Major surgery or significant traumatic injury < 28 days prior to enrollment (excluding biopsies) or anticipation of the need for major surgery during study treatment
* Clinically significant toxicities from prior treatment have not resolved to Grade </= 1 (per US national cancer institute (NCI) common terminology criteria for adverse events (CTCAE) v5.0) prior to the first study drug administration with exceptions defined by the protocol
* Evidence of any significant, concomitant disease (e.g. cardiovascular, pulmonary, liver, CVA or stroke, ILD, PML, infection, HLH etc) that could affect compliance with the protocol or interpretation of results
* For participants enrolled into glofitamab cohort: documented refractoriness to an obinutuzumab monotherapy-containing regimen (defined as disease that did not achieve response (PR or CR) or progressed within 6 months of the last dose of an obinutuzumab-containing regimen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2029-09-15 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with dose-limiting toxicities (DLTs) [dose escalation] | Until 90 days after the final dose of study treatment
Percentage of participants with adverse events [all cohorts] | Until 90 days after the final dose of study treatment
Best overall response rate (ORR), defined as the proportion of participants whose best overall response is a partial response (PR) or a complete response (CR) during the study, as determined by the investigator using Lugano 2014 criteria [dose expansion] | Up to 2 years after start of primary study treatment
Tolerability, as assessed by the incidence of dose interruptions, dose reductions, dose intensity, and treatment discontinuation [dose escalation] | Until 90 days after the final dose of study treatment

SECONDARY OUTCOMES:
Best CR rate, defined as the proportion of participants whose best overall response is a CR during the study, as determined by the investigator using Lugano 2014 criteria [all cohorts] | Up to 1 year after primary study treatment
Best ORR (CR or PR at any time) on study as determined by the investigator using Lugano 2014 criteria [dose escalation] | Up to 2 years after primary study treatment
Duration of response (DOR) as determined by the investigator using Lugano 2014 criteria [all cohorts] | Up to 2 years after primary study treatment
Progression-free survival (PFS) as determined by the investigator using Lugano 2014 criteria [dose expansion] | Up to 2 years after primary study treatment
Event-free survival (EFS) as determined by the investigator using Lugano 2014 criteria [dose expansion] | Up to 2 years after primary study treatment
Overall survival (OS) [dose expansion] | Up to 2 years after primary study treatment
Percentage of participants with adverse events [dose expansion] | Until 90 days after the final dose of study treatment
Serum concentration of subcutaneous (SC) mosunetuzumab [all cohorts] | Up to 2 years after primary study treatment
Serum concentration of intravenous (IV) glofitamab [all cohorts] | Up to 2 years after primary study treatment
Serum concentration of CC-220 and CC-99282 (CELMoDs) [all cohorts] | Up to 12 cycles of study treatment (cycle length = 21 or 28 days for Arm 1 and 21 days for Arm 2)
Tolerability, as assessed by the incidence of dose interruptions, dose reductions, dose intensity, and treatment discontinuation [dose expansion] | Until 90 days after the final dose of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (6):
  - UCSF/Hematology, Blood & Marrow Transplant, And Cellular Therapy (HBC) Program, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Chicago, Chicago, Illinois
  - Levine Cancer Institute, Charlotte, North Carolina
  - UT MD Anderson Cancer Center, Houston, Texas
- Israel (5):
  - Soroka, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Center Hospital, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (5):
  - IRCCS Azienda Ospedaliero Universitaria di Bologna, Bologna, Emilia-Romagna
  - IRCCS Istituto Romagnolo per lo studio dei tumori "Dino Amadori", Meldola, Emilia-Romagna
  - ASST Spedali Civili di Brescia, Brescia, Lombardy
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Pisana-Ospedale Santa Chia, Pisa, Piedmont
- Spain (6):
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario La Fe, Valencia, Valencia
  - Hospital Universitari Vall d Hebron, Barcelona
  - Clinica Universidad de Navarra-Madrid, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hosp Universitario Salamanca, Salamanca
- United Kingdom (4):
  - NHS Greater Glasgow and Clyde, Glasgow
  - University College London Hospitals, London
  - Nottingham University Hospitals City Campus, Nottingham
  - Oxford University Hospitals NHS Trust;Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No